CLINICAL TRIAL: NCT05528679
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II, Efficacy and Safety Study of Recombinant Anti-IL-5 Humanized Monoclonal Antibody Therapy in Adult Subjects With Severe Eosinophilic Asthma
Brief Title: A Phase II Study of 610 in Participants With Severe Eosinophilic Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-610-BA-II-01
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Asthma
Keywords: Asthma; Eosinophilic asthma; Exacerbations; 610; Placebo
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): 610 100 mg administered subcutaneously every 4 weeks
  Interventions: Drug: 610 100mg
- Treatment group B (Experimental): 610 300 mg administered subcutaneously every 4 weeks
  Interventions: Drug: 610 300mg
- placebo Arm Type：no inter (Placebo Comparator): placebo administered subcutaneously every 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 610 100mg — 100mg administered subcutaneously Q4W
  Arms: Treatment group A
Drug: 610 300mg — 300mg administered subcutaneously Q4W
  Arms: Treatment group B
Drug: placebo — administered subcutaneously Q4W
  Arms: placebo Arm Type：no inter

SUMMARY:
This study will assess the efficacy and safety of 610 as an adjunctive therapy in adult subjects with severe eosinophilic asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of 610 in adults with severe eosinophilic asthma. Plan to recruit 120 subjects, and the subjects divided into 3 groups: 610 100mg group, 610 300mg group and placebo group. The study is divided into screening period of 4 weeks, treatment period of 16 weeks and follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and follow the protocol requirements, and give written informed consent prior to participation voluntarily in the study
* Female and male aged 18 to 75 years
* Diagnosed with asthma for ≥12 months that meet GINA
* Within 6 months before screening, treatment with medium to high dose inhaled corticosteroid（ICS，inhaled fluticasone at a dosage of at least 500 μg, or equivalent, daily. ICS can be included in In the ICS/LABA combination preparation）and at least one other additional controller medication, such as long-acting β₂ receptor agonist (LABA), leukotriene receptor antagonist (LTRA), theophylline, long-acting Anticholinergic drugs (LAMA), etc. Those medicine must be stable for ≥ 28 days prior to screening and baseline and must continue without dosage changes throughout the study
* Current treatment with maintenance oral corticosteroids (OCS), prednisone dosage must be ≤10 mg, or equivalent, daily, and stable for ≥ 28 days prior to screening and baseline and must continue without dosage changes throughout the study
* In the past 12 months prior to screening， two or more asthma exacerbations history, or at least one time emergency department (ED) visits and/or ICU and/or hospitalization
* Pre-bronchodilator FEV1 <80% predicted value
* Positive of bronchodilator test or positive of bronchial provocation test
* Asthma Control Questionnaire score ≥1.5
* Asthma-related blood eosinophils ≥ 300 cells/μL within 6 months before screening, or asthma-related blood eosinophils ≥ 150 cells/μL at screening
* Male and their partners or female must commit to correct use of one or more effective contraceptive measures of the duration of the trial and for 6 months after the last study drug administration. No fertility, sperm donation, or egg donation plans for at least 6 months after the last study drug administration

Exclusion Criteria:

* With clinically important lung diseases other than asthma that may affect safety or efficacy and evaluated by investigator. This includes lung infection, chronic obstructive pulmonary disease, bronchiectasis, hypersensitivity pneumonitis, pulmonary fibrosis, Allergic bronchopulmonary aspergillosis, etc.
* With other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, eosinophilic granulomatosis with polyangiitis (EGPA), or eosinophilic esophagitis
* In past 12 months prior to screening，patients has done bronchial thermoplasty or radiotherapy or plan to do it during of the trial
* with severe cardiac disease or uncontrolled or severe cardiac arrhythmia
* poorly controlled systemic disease
* Active infection that requiring systemic treatment at screening
* Parasitic infection without adequate treatment within 6 months before screening
* Lymphoproliferative disease or any malignancy history within past 5 years prior to screening (Except for received treatment and no recurrence in the past 3 months include basal cell carcinoma, actinic keratosis, carcinoma in situ of cervix, or resected non-invasive malignant colonic polyps.)
* Liver function meets one of the following criteria at screening or before randomization: a) Serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) ≥ 2.0×ULN (upper limit of normal); b) Total bilirubin≥1.5×ULN
* At screening, HBsAg or HCV Ab or HIV Ab or TP Ab positive; HBsAg or HCV Ab positive need to be further tested of HBV DNA titer detection or HCV RNA detection (More than normal value range needs to be excluded)
* Subjects who have received any monoclonal antibody treatment within 3 months or 5 half-lives (whichever is longer) before screening, or with poor treatment effect of anti-IL-5/5R
* Vaccination history with live vaccines (including live attenuated vaccines) within 4 weeks before screening, or plan to receive during of the trial
* Participated in any interventional clinical trial and received intervention within 3 months before screening
* Allergy/intolerance to investigational medicinal product.
* Current smokers with average monthly smoking of ≥10 cigarettes within 6 months before screening, or former smokers with a smoking history of ≥10 pack years (number of pack years = (number of cigarettes per day / 20) x number of years smoked)
* Plan to pregnant during of the trial or pregnant or breastfeeding
* Any other things that are not suitable for participating in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) at week 16 | Baseline (Day 1) and at week 16
  FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry.

SECONDARY OUTCOMES:
Changes from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) at weeks 4, 8, and 12 | Baseline (Day 1) and at week 4,8,12
  FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry.
Percentage change from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) at weeks 4, 8, 12, 16 | Baseline (Day 1) and at week 4,8,12
  Percentage of FEV1 will be measured using spirometry.
Number of asthma exacerbation through study week 16 | From baseline (Day 1) to week 16
  Asthma exacerbation are defined as worsening of asthma which required use of systemic corticosteroids (≥3 days. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visits.
Time to first asthma exacerbation event | From baseline (Day 1) to week 16
  Asthma exacerbation are defined as worsening of asthma which required use of systemic corticosteroids (≥3 days. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visits.
Number of asthma exacerbations requiring hospitalization (including intubation and ICU admission) or emergency room visits (not conversion to hospitalization) | From baseline (Day 1) to week 16
  Asthma exacerbations that are associated with a hospitalization or an emergency room visit.
Number of asthma exacerbations requiring hospitalization (including intubation and ICU admission) | From baseline (Day 1) to week 16
  Asthma exacerbations that are associated with a hospitalization.
Puffs of rescue medication for asthma exacerbations | From baseline (Day 1) to week 16
  Albuterol or levalbuterol for an asthma exacerbation is considered rescue medication.
Change from baseline in Asthma Control Questionnaire score at week 4,8,12,16 | Baseline (Day 1) and at week 4,8,12,16
  The ACQ has 7 questions- the first 5 items assess the most common asthma symptoms plus 6. short-acting bronchodilator use and 7. FEV1 (pre-bronchodilator use, % and % predicted use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6= maximum impairment).
Change From Baseline in the St. George's Respiratory Questionnaire Total Score at week 16 | Baseline (Day 1) and at week 16
  The St. George's Respiratory Questionnaire is an established instrument, comprising 50 questions, evaluating symptoms, activity, and impacts; to measure Quality of Life in participants with diseases of airway obstruction and to elicit the participant's opinion of his/her health.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghong Zhou, MD, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.; Min Zhang, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Xin Zhou, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided